CLINICAL TRIAL: NCT05460637
Title: Physical Activity Intervention Tailored for Rural Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacob Gallagher (Other)
Collaborators: Iowa State Fraternal Order of Eagles (Unknown)
Responsible Party: Sponsor-Investigator, Jacob Gallagher, Graduate Fellow, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 202201021
Record Dates: First submitted 2022-07-07; First posted 2022-07-15 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Physical Inactivity; Sedentary Behavior; Weak; Muscle
Keywords: physical activity; sedentary behavior; strength training; mHealth; rural; scalable
MeSH Terms: conditions — Sedentary Behavior; Asthenia; Motor Activity

STUDY DESIGN:
Intervention Model Description: This study uses a single-arm study with all participants receiving the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Participants receive a Fitbit and access to a 10 week educational course that accessible through the web or app. While participants can complete the program at their own pace, there is a suggested schedule with 1-2 modules/lessons completed per week. Each module has a different topic related to promoting adoption and maintenance of physical activity.
  Interventions: Behavioral: No BS just Fitness

INTERVENTIONS:
Behavioral: No BS just Fitness — The participants receive lessons on the physical activity guidelines, goal setting, physical activity planning, habit development, identity formation, and how to apply all these tools together. In addition, there are numerous resources provided to other existing web resources, including exercise videos and other informational webpages (e.g., USDA nutritional recommendations).

SUMMARY:
The goal of this project is to develop a scalable physical activity intervention tailored to rural men. We will recruit participants nationwide from ResearchMatch data base, emails, and social media posts. Participants will have access to health education materials hosted on Healthie, a health coaching software platform, and provided an activity monitor (e.g., Fitbit) to support behavior change. The health education materials provide participants with education, motivation, and support for making health behavior change (e.g., increasing physical activity levels). We will measure physical activity behaviors, psychosocial, and several health outcomes

ELIGIBILITY:
Inclusion Criteria:

* Have a smart phone capable of sending/receiving test messages
* Currently inactive (<75 minutes of moderate-vigorous activity per week)
* Identify as male
* Live in a rural community
* Intending to be more active

Exclusion Criteria:

* Not able to safely increase physical activity
* Cannot commit to a 10 week program
* Have a surgery planned in 6 months

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — We are asking participants to select what gender best describes them. Since our program is tailored specifically to the needs of men, we are recruiting only participants who identify as males.
Enrollment: 40 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Physical Activity (average steps per day) | Measurements taken from Baseline (Week 0) to post-intervention (Week 11)
  Examining the activity levels of participants using the average steps per day from the Fitbit device. The average steps per day taken during baseline (Week 0) will be compared to average steps per day during post-intervention testing (Week 11).

SECONDARY OUTCOMES:
Muscular Strength | Measurements taken from Baseline (Week 0) to post-intervention (Week 11)
  Assessed via a sum score of push-ups (until exhaustion), squat test (number of reps in 60s), and sit-up (reps in 60s)
Attitude towards physical activity (self-report) | Measurements taken at Baseline (Week 0) and at post-intervention (Week 11)
  Attitude towards physical activity will be measured using a sum score of Likert scales (1- Extremely disagree to 7-Extremely agree) on 6 questions, asking about participants' belief regarding physical activity (e.g., engaging in physical activity would be enjoyable) - (Rhodes & Courneya, 2003).
Perceived capability over physical activity (self-reported) | Measurements taken at Baseline (Week 0) and at post-intervention (Week 11)
  Perceived capability over physical activity will measured using a sum score of Likert scales (1- Extremely disagree to 7-Extremely agree) on 3 questions, asking about participants' confidence over engaging in physical activity (e.g., I possess the skill to do regular physical activity if I wanted to) (Rhodes, Blanchard, & Matheson, 2006; Burrell, Allan, Williams, & Jonnston, 2018)
Perceived opportunity for physical activity (self-reported) | Measurements taken at Baseline (Week 0) and at post-intervention (Week 11)
  Perceived opportunity for physical activity will be measured using a sum score of Likert scales (1- Extremely disagree to 7-Extremely agree) on 3 questions, asking about participants' opportunity to engage in physical activity (e.g., If I really wanted to do regular physical activity, I would have the chance to do so) (Rhodes, Blanchard, & Matheson, 2006; Burrell, Allan, Williams, & Jonnston, 2018)
Behavioral regulation for physical activity (self-reported) | Measurements taken at Baseline (Week 0) and at post-intervention (Week 11)
  Behavioral regulation for physical activity will be measured using a sum score of Likert scales (1- Extremely disagree to 7-Extremely agree) on 6 questions, asking about participants' strategies used to help them engage in physical activity (e.g., I kept track of my physical activity in a dairy or log over the last month) (Sniehotta, Schwarzer, Scholz, & Shuz, 2005)
Habit of physical activity (self-reported) | Measurements taken at Baseline (Week 0) and at post-intervention (Week 11)
  Habit of physical activity will be measured as a sum score of Likert scales (1- Extremely disagree to 7-Extremely agree) on 4 questions, asking about participants' habits related to physical activity (e.g., Physical activity is something I do automatically) (Gardner, Abraham, Lally, de Brujin, 2012))
Physical activity identity (self-reported) | Measurements taken at Baseline (Week 0) and at post-intervention (Week 11)
  Physical activity identity will be measured as a sum score of Likert scales (1- Extremely disagree to 7-Extremely agree) on 4 questions, asking about participants' personal beliefs about their identity and physical activity (e.g., I consider myself someone who does regular physical activity) (Wilson & Muon, 2008; Sparks & Shepard, 1992)
Decisional Intentions to be physically active (self-reported) | Measurements taken at Baseline (Week 0) and at post-intervention (Week 11)
  Participants will be asked to fill in the blank: "I intend to engage in physical activity ______ times this next week" with the number of days they intend to be active. (Courneya, 1994)

CONTACTS AND LOCATIONS:
Locations (1):
- Field House, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
All data related to the primary outcome will be shared.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The data will become available within 6 months after related publications.
Access Criteria: Data will be made available using a repository at the University of Iowa. This data will be available to use for replication of results, and secondary analysis.

DOCUMENTS (1):
  • Informed Consent Form (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT05460637/ICF_000.pdf